CLINICAL TRIAL: NCT03942224
Title: A Randomized Phase II Study of DaRatumumab, Ixazomib, and Dexamethasone vs Daratumumab, Bortezomib (VElcade) and Dexamethasone Followed by Daratumumab-Ixazomib-Dexamethasone in Newly Diagnosed Multiple Myeloma (DeRIVE Study)
Brief Title: Daratumumab, Ixazomib, & Dexamethasone or Daratumumab, Bortezomib, & Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma
Acronym: DeRIVE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Takeda (Industry); Janssen, LP (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Nooka, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00102336; NCI-2018-03615 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4547-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; daratumumab; Antibodies, Monoclonal; Dexamethasone; Calcium Dobesilate; ixazomib; MLN2238

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (DId) (Experimental): INDUCTION: Patients receive dexamethasone IV and PO on days 1, 8, 15, and 22, daratumumab IV on days 1, 8, 15, and 22 of cycles 1-2 and on days 1 and 15 of cycles 3-8, and ixazomib PO on days 1, 8, and 15. Treatment repeats every 28 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Eligible patients then undergo stem cell transplant per standard of care. Patients who have at least stable disease after induction and patients who have undergone transplant continue to Maintenance.
  MAINTENANCE: Patients receive dexamethasone IV and PO on days 1, 8, 15, and 22, daratumumab IV on day 1, and ixazomib PO on days 1, 8, and 15. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab; Drug: Dexamethasone; Drug: Ixazomib
- Arm II (DVd, DId) (Experimental): INDUCTION CYCLES 1-3: Patients receive dexamethasone IV and PO on days 1, 8, and 15, daratumumab IV on days 1, 8, and 15, and bortezomib subcutaneously (SC) on days 1, 4, 8, and 11. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity.
  INDUCTION CYCLES 4-8: Patients receive dexamethasone IV and PO on days 1, 8, 15, and 22, daratumumab IV on days 1 and 15, and ixazomib PO on days 1, 8, and 15. Treatment repeats every 28 days for 5 cycles in the absence of disease progression or unacceptable toxicity. Eligible patients then undergo stem cell transplant per standard of care. Patients who have at least stable disease after induction and patients who have undergone transplant continue to Maintenance.
  MAINTENANCE: Patients receive dexamethasone IV on day 1, daratumumab IV on day 1, and ixazomib PO on days 1, 8, and 15. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Biological: Daratumumab; Drug: Dexamethasone; Drug: Ixazomib

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: MLN341; PS-341; Velcade
  Arms: Arm II (DVd, DId)
Biological: Daratumumab — Given IV
  Other Names: Anti-cluster of differentiation 38 (CD38) Monoclonal Antibody; Darzalex; HuMax-CD38
Drug: Dexamethasone — Given IV and PO
  Other Names: Decadron; Dexasone; Diodex; Hexadrol; Maxidex
Drug: Ixazomib — Given PO
  Other Names: Ninlaro; MLN2238

SUMMARY:
This phase II trial studies how well daratumumab, ixazomib, and dexamethasone with or without bortezomib work in treating patients with newly diagnosed multiple myeloma. Immunotherapy with monoclonal antibodies, such as daratumumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as ixazomib, dexamethasone, and bortezomib, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving daratumumab, ixazomib, and dexamethasone with or without bortezomib may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the ≥ very good partial response (VGPR) rate after 8 cycles in subjects treated with daratumumab, ixazomib and dexamethasone (DId) versus (vs) daratumumab, bortezomib and dexamethasone (DVd) followed by DId among newly diagnosed myeloma patients (NDMM).

SECONDARY OBJECTIVES:

I. To estimate the proportion of subjects with successful stem cell mobilization after receiving 3 cycles of treatment in both arms (DId x 8 vs DVd x 3 then DId x 5).

II. To establish safety among patients receiving the combination of DId and DVd then DId.

III. To obtain anti-tumor activity (best response rates: overall response rate [ORR], VGPR, complete response [CR], stringent complete response [sCR] and minimal residual of disease [MRD] negativity) in patients treated with these combinations.

IV. Progression free survival (PFS), progression free survival 2 (PFS2), duration of response (DOR), time to progression (TTP), determine the time to next therapy (TTNT).

V. Overall survival (OS).

VI. Engraftment parameters among the autologous stem cell transplant (ASCT) group.

VII. Determine whether tumor response and PFS may change in subgroups with different prognosis according to current prognostic factors.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I:

INDUCTION: Patients receive dexamethasone intravenously (IV) and orally (PO) on days 1, 8, 15, and 22, daratumumab IV on days 1, 8, 15, and 22 of cycles 1-2 and on days 1 and 15 of cycles 3-8, and ixazomib PO on days 1, 8, and 15. Treatment repeats every 28 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Eligible patients then undergo stem cell transplant per standard of care. Patients who have at least stable disease after induction and patients who have undergone transplant continue to Maintenance.

MAINTENANCE: Patients receive dexamethasone IV and PO on days 1, 8, 15, and 22, daratumumab IV on day 1, and ixazomib PO on days 1, 8, and 15. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

ARM II:

INDUCTION CYCLES 1-3: Patients receive dexamethasone IV and PO on days 1, 8, and 15, daratumumab IV on days 1, 8, and 15, and bortezomib subcutaneously (SC) on days 1, 4, 8, and 11. Treatment repeats every 21 days for 3 cycles in the absence of disease progression or unacceptable toxicity.

INDUCTION CYCLES 4-8: Patients receive dexamethasone IV and PO on days 1, 8, 15, and 22, daratumumab IV on days 1 and 15, and ixazomib PO on days 1, 8, and 15. Treatment repeats every 28 days for 5 cycles in the absence of disease progression or unacceptable toxicity. Eligible patients then undergo stem cell transplant per standard of care. Patients who have at least stable disease after induction and patients who have undergone transplant continue to Maintenance.

MAINTENANCE: Patients receive dexamethasone IV on day 1, daratumumab IV on day 1, and ixazomib PO on days 1, 8, and 15. Cycles repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria on screening examination to be eligible to participate in the study. All laboratory assessments should be performed within 21 days of initiation of protocol therapy unless otherwise specified. Subject is, in the investigator's opinion, willing and able to comply with the protocol requirements
* Subject has given voluntary signed written informed consent before performance of any study-related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to their future medical care
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Have documented multiple myeloma as defined by the International Myeloma Working Group (IMWG) 2014 criteria including: Clonal bone marrow plasma cells ≥ 10% (If bone marrow has less than 10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement). In addition, the patient must meet one of the criteria in d1 or d2:

  * Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically (one or more of the following):

    * Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal (ULN) or > 2.75 mmol/L (> 11 mg/dL)
    * Renal insufficiency: Creatinine clearance (CrCl) < 40 mL/min (measured or estimated by validated equations) or serum creatinine > 177 umol/L (> 2 mg/dL)
    * Anemia: hemoglobin value of > 20 g/L below the lower limit of normal, or a hemoglobin value < 100 g/L
    * Bone lesions: 1 or more osteolytic lesions on skeletal radiography, computed tomography (CT), or magnetic resonance imaging (MRI)

      * Clonality should be established by showing kappa/lambda-light-chain restriction on flow cytometry, immunohistochemistry, or immunofluorescence. Bone marrow plasma cell percentage should preferably be estimated from a core biopsy specimen; in case of a disparity between the aspirate and core biopsy, the highest value should be used
  * Any one or more of the following:

    * Clonal bone marrow plasma cell percentage ≥ 60%

      * Clonality should be established by showing kappa/lambda-light-chain restriction on flow cytometry, immunohistochemistry, or immunofluorescence. Bone marrow plasma cell percentage should preferably be estimated from a core biopsy specimen; in case of a disparity between the aspirate and core biopsy, the highest value should be used
    * Involved:uninvolved serum free light chain (FLC) ratio > 100

      * These values are based on the serum Freelite assay (The Binding Site Group, Birmingham, UK). The involved FLC must be ≥ 100 mg/L
    * > 1 focal lesions on MRI studies; Each focal lesion must be 5 mm or more in size
* Measurable disease as defined by any of the following:

  * Serum M-protein level ≥ 1.0 g/dL or urine M-protein level ≥ 200 mg/24 hours. Note: All attempts should be made to determine eligibility of the subject based on the central laboratory results of screening blood and urine M-protein measurements. In exceptional circumstances, the local laboratory results for blood and urine M-protein measurements may be used to determine eligibility, but only if the results are clearly (eg, 25% or more) above the thresholds for measurability; or
  * Immunoglobulin A (IgA), immunoglobulin D (IgD), immunoglobulin E (IgE), or immunoglobulin M (IgM) multiple myeloma: serum M-protein level ≥ 0.5 g/dL or urine M-protein level ≥ 200 mg/24 hours; or
  * Light chain multiple myeloma without measurable disease in the urine: serum Ig FLC ≥ 10 mg/dL and abnormal serum Ig kappa/lambda FLC ratio
* Prior treatment to stabilize the patient with steroids up to 160 mg IV equivalents of dexamethasone is allowed
* Prior treatment to stabilize the patient with bortezomib up to 2 doses of 1.3 mg/m² each dosing equivalent is allowed
* Subject agrees to refrain from blood donations during therapy on study and for 8 weeks after therapy is completed
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
  * Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-International Unit (mIU)/mL within 10-14 days prior to and again within 24 hours of starting study drugs
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

* Diagnosed with smoldering multiple myeloma (MM), monoclonal gammopathy of undetermined significance, Waldenstrom's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome, amyloidosis or primary or secondary plasma cell leukemia
* Participant has ≥ grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination within 21 days before initiation of protocol therapy
* Renal insufficiency, defined as creatinine clearance ≤ 30 mL/min (either actual or calculated value), within 21 days of initiation of protocol therapy. The Cockcroft-Gault formula should be used for calculating creatinine clearance values
* Platelet count ≤ 75,000 cells/mm³ at time of screening evaluation. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment
* Participants with an absolute neutrophil count (ANC) ≤ 1000 cells/mm³ at time of screening evaluation. Growth factors may not be used to meet ANC eligibility criteria within 14 days of obtaining screening evaluation
* Participants with hemoglobin level < 7.0 g/dL, at time of screening. Transfusion may not be used to meet eligibility criteria within 7 days of obtaining screening evaluation
* Participants with hepatic impairment, defined as bilirubin ≥ 1.5 x institutional upper limit of normal (ULN) or aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]), or alkaline phosphatase ≥ 3 x institutional ULN, within 21 days of initiation of protocol therapy
* Patients may be receiving concomitant therapy with bisphosphonates and low dose corticosteroids (e.g., prednisone up to but no more than 10 mg p.o. once daily (q.d.) or its equivalent) for symptom management and comorbid conditions. Doses of corticosteroid should be stable for at least 7 days prior to study treatment.)
* Steroids more than 160 mg IV equivalents of dexamethasone or bortezomib > 2 doses of 1.3 mg/m² each dosing equivalents
* Known significant cardiac abnormalities including:

  * Congestive heart failure, New York Heart Association (NYHA) class III or IV
  * Uncontrolled angina, arrhythmia or hypertension
  * Myocardial infarction within the past six months
  * Any other uncontrolled or severe cardiovascular condition
  * Prior cerebrovascular event with residual neurologic deficit
* Known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal
* Has known moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification
* Serious, intercurrent illness including, but not limited to, clinically relevant active infection, uncontrolled diabetes mellitus, or serious co-morbid medical conditions such as chronic restrictive pulmonary disease, and cirrhosis
* Seropositive for human immunodeficiency virus (HIV)
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
* Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)
* Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Known hypersensitivity to acyclovir or similar anti-viral drug
* Known intolerance to steroid therapy
* Participants with known central nervous system (CNS) involvement
* Poor tolerability or known allergy to any of the study drugs or compounds of similar chemical or biologic composition to dexamethasone, boron or mannitol
* Female participants pregnant or breast-feeding
* Participants who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of the surgery
* Participants with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff
* Prior exposure to anti-CD38 therapy
* Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong cytochrome P450, family 3, subfamily A (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial
* Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
≥ Very good partial response (VGPR) response rate | After cycle 8 (224 days)
  This will be defined as the proportion of subjects who achieved a response of VGPR or better (stringent complete response [sCR], complete response [CR], or VGPR) after induction cycle 8 treatment. Response will be determined by modified International Myeloma Working Group (IMWG) criteria.

SECONDARY OUTCOMES:
Stem cell mobilization | After cycle 3 (84 days)
  This will be defined as the proportion of subjects with successful stem cell mobilization after induction cycle 3. A successful stem cell mobilization is defined as the ability to collect a total of at least 2 x 10⁶ cluster of differentiation 34+ (CD34+) cells/kg.
Best response on study | Up to 5 years after study start
  Best response on study refers to the best response prior to discontinuation of all study therapy.
Objective response rate (ORR) | Up to 5 years after study start
  Objective response rate will be defined as the proportion of treated subjects who achieve a best response of CR, sCR, VGPR, or partial response (PR) using the IMWG criteria.
Minimal residual disease (MRD) | Up to 5 years after study start
  The achievement of minimal residual disease will be evaluated and reported on patients that achieve a complete response. Next-Generation sequencing will be performed to evaluate MRD.
Progression-Free Survival (PFS) | Up to 5 years after study start
  Progression-free survival (PFS) is defined as the time from first dose of study drug until documented progression or death. A subject who neither progresses nor dies will be censored on the date of his or her last tumor assessments.
Time to response | Up to 5 years after study start
  Time to response is defined as the time from first dose of study drug to the first documentation of response PR or better. This analysis will be restricted to subjects whose best response is PR or better.
Duration of response (DOR) | Up to 5 years after study start
  Duration of response is the time from first response (PR or better) until a progression event (documented progression or death). Only subjects who ever achieved a response of PR or better will be considered. Subjects who neither progress nor die will be censored on the date of their last tumor assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Nooka, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/24/NCT03942224/ICF_000.pdf